CLINICAL TRIAL: NCT02055794
Title: Promoting Optimal Healing After Laceration Repair Study - PALS Study
Brief Title: Promoting Optimal Healing After Laceration Repair Study
Acronym: PALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Dee Fenner, Professor, Obstetrics & Gynecology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00079230
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Neuralgia, Perineal
Keywords: perineal wound; perineal tear; perineum; pain; childbirth
MeSH Terms: conditions — Neuralgia; Pain | interventions — Enbucrilate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Suturing of the perineal skin (Active Comparator): Suturing of the perineal skin after deep vaginal and perineal tissues are closed using a continuous 3-0 Vicryl suture.
  Interventions: Procedure: Suturing of the perineal skin
- No suturing of the perineal skin (Active Comparator): No suturing of the perineal skin after deep vaginal and perineal tissues are closed using a continuous 3-0 Vicryl suture.
  Interventions: Procedure: No suturing of the perineal skin
- Closing perineal skin with surgical glue (Active Comparator): Closure of the perineal skin with n-Butyl 2-cyanoacrylate (Indermil®) surgical glue after deep vaginal and perineal tissues are closed using a continuous 3-0 Vicryl suture.
  Interventions: Procedure: Closing perineal skin with surgical glue

INTERVENTIONS:
Procedure: Suturing of the perineal skin
  Arms: Suturing of the perineal skin
Procedure: Closing perineal skin with surgical glue
  Other Names: n-Butyl 2-cyanoacrylate; Indermil®; surgical glue
  Arms: Closing perineal skin with surgical glue
Procedure: No suturing of the perineal skin
  Arms: No suturing of the perineal skin

SUMMARY:
The goal of this research is to investigate three different methods of perineal skin closure during second-degree perineal wound repair and determine which method is associated with the least amount of patient pain.

Null hypothesis: There will be no difference in patient pain among the three different methods for second degree perineal wound repair.

DETAILED DESCRIPTION:
At the University of Michigan, there are currently two standard techniques for repairing second-degree perineal lacerations that differ only in management of the perineal skin :

1. Closure of the deep tissues and superficial perineal skin using a continuous 3-0 Vicryl suture
2. Closure of the deep tissues with a continuous 3-0 Vicryl suture and reapproximation of, but not suture-closure of the perineal skin.

The primary goal of our study is to compare patient pain amongst the following three perineal skin repair techniques after second degree laceration:

1. Perineal skin closure with suturing
2. Not suturing the perineal skin
3. Closure of the perineal skin with n-Butyl 2-cyanoacrylate (Indermil®) surgical glue.

In all women, the deep vaginal and perineal tissues will be closed using a continuous 3-0 Vicryl suture, as is current standard practice.

Aim: To assess and compare patient pain among the three groups at intervals of 1 day, 2 weeks, 6 weeks and 3 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years old - 45 years old
* Immediately post-vaginal birth, including forceps-assisted vaginal delivery, vacuum-assisted vaginal delivery
* > 32 weeks gestation
* Second degree laceration from spontaneous tear or midline episiotomy
* Proficient in English

Exclusion Criteria:

* <18 years old and >45 years old
* Delivery by Cesarean
* 1st, 3rd or 4th degree lacerations
* Induction for intrauterine fetal demise or terminal fetal condition, or any instance where immediate status of the newborn is unknown
* Known allergy to cyanoacrylate or formaldehyde
* Systemic infections, uncontrolled diabetes (women with well-controlled pre-gestational or gestational diabetes will not be excluded)
* History of connective tissue disorders (e.g. Scleroderma, Ehlers Danlos)
* Chronic use of steroids
* Currently under treatment for cancer
* Previous radiation to the pelvis
* Any organ transplants
* History of neurological conditions including multiple sclerosis, stroke, Alzheimer's, or other dementias
* Not proficient in the English language

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Patient-perceived pain | Post-partum (PPD), 2 weeks, 6 weeks and 3 months.
  The 2 week and 3 month measurements will be done via email, web or mailed questionnaire. Pain will be measured using 3 pain scales: a validated 100-mm Visual Analogue Scale (VAS) (anchors: 0 = none, 100 mm = worst imaginable), a 6 point Likert scale and the McGill pain questionnaire short form.

SECONDARY OUTCOMES:
Wound assessment | 6 weeks post-partum
  Wounds will be assessed through wound evaluation (6 weeks post-partum), wound complications (wound infection, dehiscence, granulation tissue), need for additional interventions (silver nitrate, revision of wound) and assessment of wound appearance using a validated 100-mm VAS (anchors: 0 = worst scar, 100 mm = best scar).

CONTACTS AND LOCATIONS:
Overall Officials: Dee Fenner, M.D., Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No